CLINICAL TRIAL: NCT04883606
Title: Non-interventional, Multicenter Retrospective Study of the Effectiveness and Safety of Teduglutide (Revestive®) in Short Bowel Syndrome Adult Patients in Spain (T-Rex Study)
Brief Title: A Study With Teduglutide (Revestive®) in Adults With Short Bowl Syndrome
Acronym: T-Rex
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-4002; MACS-2020-04220 (Other: Takeda)
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Retrospective data will be collected from participants who followed up at least 6 months before teduglutide initiation or intestinal failure associated with SBS-IF diagnosis and at least 6 months of follow-up after teduglutide treatment initiation.

SUMMARY:
The main aims of the study are to assess the safety profile of teduglutide (Revestive®) as well as how many people with Short Bowl Syndrome experience a reduction of parenteral support when treated with teduglutide (Revestive®).

This study is about collecting existing data only; participants will not receive teduglutide (Revestive®) as part of this study. No new information will be collected during this study. Only data already available in the hospital records will be reviewed and collected for this study.

Participants do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants >= 18 years of age diagnosed with intestinal failure due to SBS as a result of intestinal resection.
* SBS-IF participants treated with teduglutide according to Summary of Product Characteristics (SmPC).
* Patients who receive or have received teduglutide for at least six months at the date of inclusion (from treatment initiation to inclusion date, date of discontinuation, death for any cause or loss of follow-up).
* When required by the ethics committee of the center: participants who have signed the informed consent form (ICF) to participate in the study.

Exclusion Criteria:

- Participants who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SBS-IF participants with age greater than equal to (>=) 18 years treated with teduglutide in Spain.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Response of 20 Percent (%) to 100% Reduction From Baseline in Weekly Parenteral Support (PS) Volume at Month 1 | Month 1
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 1 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 2 | Month 2
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 2 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 3 | Month 3
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 3 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 6 | Month 6
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 6 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 9 | Month 9
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 9 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 12 | Month 12
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 12 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 18 | Month 18
  Percentage of participants achieveing response of 20% to 100% reduction from baseline in weekly PS volume at Month 18 after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume at Month 24 | Month 24
  Percentage of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume at Month 24 after teduglutide treatment initiation will be reported.

SECONDARY OUTCOMES:
Average Change in Weekly Volume of Parenteral Nutrition (PN)/Intravenous (IV) Requirement | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in weekly volume of PN/IV requirement since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Time to Achieve Response up to Month 24 | Baseline up to Month 24
  Response is defined as the achievement of a 20% to 100% reduction in weekly PS volume from baseline up to Month 24.
Average Change in PN/IV Caloric Intake | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in PN/IV calories intake since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Average Change in Number of Days per Week With PN/IV Usage | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in number of days per week with PN/IV since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Number of Participants Achieving Response of 20% to 100% Reduction From Baseline in Weekly PS Volume | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Number of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume since 6 months before teduglutide treatment initiation to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be reported.
Number of Participants With Independence From PN and IV Fluid Support | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Number of participants with independence from PN and IV fluid support since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Median Time to Achieve any Response After Teduglutide Treatment Initiation. | Up to Month 24
  Median time to achieve any response after teduglutide treatment initiation will be assessed.
Median Time to Achieve Independence From PN and IV Fluid Support | Up to Month 24
  Median time to achieve independence on PN and IV fluid support after treatment with teduglutide will be assessed.
Average Change in Body Mass Index (BMI) | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in BMI after treatment with teduglutide since 6 months before teduglutide treatment initiation up to 1, 2, 3, 6, 9, 12, 18 and 24 months after teduglutide treatment initiation will be assessed.
Average Change in Daily Urine Volume | 6 months before teduglutide treatment initiation up to Months 1, 2, and 3 after teduglutide treatment initiation
  Average change in daily urine volume since 6 months before teduglutide treatment initiation up to Months 1, 2, and 3 after teduglutide treatment initiation will be assessed.
Average Change in Stool Characteristics | 6 months before teduglutide treatment initiation up to Month 6 after teduglutide treatment initiation
  Average change in stool characteristics from 6 months before teduglutide treatment initiation up to Month 6 after teduglutide treatment initiation will be assessed.
Average Change in Daily Fluids Intake | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in fluids daily intake since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Average Change in Daily Calories Oral Intake | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in daily calories oral intake since 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation will be assessed.
Average Change in Blood Parameters Such as Serum Albumin and Serum Pre-albumin | 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 9, 12, 18 and 24 after teduglutide treatment initiation
  Average change in blood parameters such as serum albumin and serum pre-albumin will be analyzed at 6 months before teduglutide treatment initiation up to Months 1, 2, 3, 6, 12, 18 and 24 after teduglutide treatment initiation.
Number of Participants With Adverse Events (AEs) | Up to Month 6 after teduglutide treatment discontinuation
  An adverse event (AEs) is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. A Serious adverse event (SAE) is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event.
Number of Participants who Discontinued Treatment due to any Cause | Up to Month 24
  Number of participants who discontinued treatment due to any cause (treatment discontinuation, worsening health conditions, withdrawal of consent) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60a511581f1122001e30a7df